CLINICAL TRIAL: NCT05082012
Title: Prospective Clinical StuDy of Tri-planar Tarsometatarsal (TMT) ArthroDesis With Early Weight-Bearing After Lapiplasty® ProceDure Through a Mini-Incision™ Approach (Mini3D)
Brief Title: Early Weight-Bearing After the Lapiplasty Mini-Incision Procedure (Mini3D)
Acronym: Mini3D
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Corporate decision to early term study to prepare for publication and addition of new studies
Sponsor: Treace Medical Concepts, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP2021-1
Record Dates: First submitted 2021-09-14; First posted 2021-10-18 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Hallux Valgus; Bunion
MeSH Terms: conditions — Hallux Valgus; Bunion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Treatment of Hallux Valgus — Patients 14 years through 58 years with symptomatic hallux valgus will be eligible to participate based on the inclusion/exclusion criteria established in the study protocol. Anticipated subject duration will be 2 years post index procedure.
  Other Names: Lapiplasty® Mini-Incision™ Procedure

SUMMARY:
Prospective, multicenter, unblinded study to evaluate outcomes of the Lapiplasty® Procedure using the Lapiplasty® Mini-Incision™ System for patients in need of hallux valgus surgery.

Up to 200 subjects will be treated in this study at up to 20 clinical sites. Patients 14 years through 58 years with symptomatic hallux valgus will be eligible to participate based on the inclusion and exclusion criteria defined in the study protocol.

DETAILED DESCRIPTION:
Prospective, multicenter, unblinded study to evaluate outcomes of the Lapiplasty® Procedure using the Lapiplasty® Mini-Incision™ System for patients in need of hallux valgus surgery:

1. To determine radiographic recurrence of hallux valgus and the timing of failure following hallux valgus correction with the Lapiplasty® Procedure.
2. To determine whether the Lapiplasty® Procedure effectively corrects anatomical alignment of the 1st metatarsal and sesamoids in all three planes.
3. To assess whether early weight-bearing after the Lapiplasty® Procedure affects the union rates or causes loss of 3-plane correction.
4. To evaluate the quality of life and pain scores following the Lapiplasty® Procedure.

ELIGIBILITY:
Inclusion Criteria:

Patients satisfying the following criteria will be considered the screening population and will be eligible for participation:

1. Male and females between the ages 14 and 58 years at the time of consent;
2. Closed physeal plates at the time of consent;
3. Intermetatarsal angle is between 10.0˚ - 22.0˚;
4. Hallux valgus angle is between 16.0˚ - 40.0˚;
5. Willing and able to adhere to early weight-bearing instructions post-operatively;
6. Capable of completing self-administered questionnaires;
7. Acceptable surgical candidate, including use of general anesthesia;
8. Female patients must be of non-child bearing potential or have a negative pregnancy test within 7 days prior to index procedure;
9. Willing and able to schedule index procedure within 3 months of consent and able to return for scheduled follow-up visits;
10. Willing and able to provide written informed consent.

Exclusion Criteria:

Patients satisfying the following criteria will not be eligible for participation:

1. Previous surgery for hallux valgus on operative side;
2. Previous surgeries on operative foot involving fusion of foot or ankle joints (other than hammertoe or lesser toes/digits);
3. Additional concomitant procedures outside of the 1st ray;
4. Moderate or Severe osteoarthritis of the MTP joint based on radiographic imaging (including lack of evident crista) or positive grind test;
5. Symptomatic flatfoot or asymptomatic flatfoot (defined as calcaneal inclination <5˚and talonavicular subluxation/uncovering >50%);
6. BMI >40 kg/m²;
7. Current nicotine user, including current use of nicotine patch;
8. Current clinical diagnosis of diabetes with fasting plasma glucose > 126 mg/dL and/or HbA1c ≥7.0;
9. Current clinical diagnosis of peripheral neuropathy or by assessment on 4-point monofilament test;
10. Current clinical diagnosis of fibromyalgia;
11. Current clinical diagnosis of Complex Regional Pain Syndrome/Reflex Sympathetic Dystrophy (CRPS/RSD);
12. Current uncontrolled hypothyroidism;
13. Previously sensitized to titanium;
14. Currently taking oral steroids or rheumatoid biologics;
15. Currently taking immunosuppressant drugs;
16. Insufficient quantity or quality of bone to permit stabilization, conditions that retard healing (not including pathological fractures) and conditions causing poor blood supply such as peripheral vascular disease;
17. Active, suspected or latent infection in the affected area;
18. Use of synthetic or allogenic bone graft substitutes;
19. Current diagnosis of metatarsus adductus (defined as MAA ≥ 23˚);
20. Known keloid and hypertrophic scar forming;
21. Scheduled to undergo a same-day bilateral procedure. Patient agrees to refrain from the Lapiplasty® Procedure (or other hallux valgus procedures) on contralateral foot for minimum of 6 months post index procedure;
22. Patient has previously been enrolled into this study for a contralateral procedure;
23. Scheduled for any concomitant procedure that would alter patient's ability to early weight-bear post-procedure;
24. Patient requires an incision >4.0 cm to complete the procedure (determined pre-operatively or intra-operatively);
25. Patient is actively involved with a workman's compensation case or is currently involved in litigation;
26. Patient is currently or has participated in a clinical study in the last 30 days prior to signing informed consent or is considering participation in another research protocol during this study. Exceptions to this include survey clinical studies with no treatment or if subject is greater than 12 months post procedure in the Treace ALIGN3D™ study without ongoing protocol defined AE; these are not exclusionary;
27. Patient has a condition or finding that, in the opinion of the Investigator, may jeopardize the patient's well-being, the soundness of this clinical study, or could interfere with provision of informed consent, completion of tests, therapy, or follow-up.

Ages: 14 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 123 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
Radiographic Recurrence | 24 months
  To determine radiographic recurrence of hallux valgus and the timing of failure following hallux valgus correction with the Lapiplasty® Procedure

SECONDARY OUTCOMES:
Radiographic Angular/Positional Alignment | pre-op, 6 weeks, 4 months, 6 months, 12 months, 24 months post Lapiplasty® Procedure
  Change in radiographic angular/positional alignment before/after the Lapiplasty® Procedure
Radiographic Healing | 12 months post Lapiplasty® Procedure
  Union vs non-union -- Non-union defined as lucency at TMT joint, hardware failure and/or loss of correction, plus clinical pain at first TMT joint
Clinical complications due to Lapiplasty® System Implants, the procedure, the post-op weight-bearing protocol or health conditions that could affect other outcome measures - measured by Adverse Events and Product Complaint data | 24 months post Lapiplasty® Procedure
  Clinical complications due to Lapiplasty® System Implants, the procedure, the post-op weight-bearing protocol or health conditions that could affect other outcome measures - measured by Adverse Events and Product Complaint data
Time to start weight-bearing in a boot | 0-3 weeks, post Lapiplasty® Procedure
  Time to start weight-bearing in a boot
Time to start weight-bearing in a shoe | 6 weeks, post Lapiplasty® Procedure
  Time to start weight-bearing in a shoe
Time to return to full unrestricted activity | 6 weeks - 6 months, post Lapiplasty® Procedure
  Time to return to full unrestricted activity
Change in Pain | 0-2 weeks, 2-3 weeks, 6 weeks, 4 months, 6 months, 12 months, 24 months post Lapiplasty® Procedure
  Change in pain assess via Visual Analog Scale (VAS)
Change in Quality of Life | 6 months, 12 months, 24 months post Lapiplasty® Procedure
  Change in quality of life via PROMIS-29, PROMIS-25, MOxFQ
Change in Range of Motion | 12 months, 24 months post Lapiplasty® Procedure
  1st MTP dorsiflexion and plantarflexion
Change in Radiographic Foot Length | 12 months post Lapiplasty® Procedure
  Change in radiographic foot length compared to baseline visit
Change in Radiographic Foot Width | 12 months post Lapiplasty® Procedure
  Change in radiographic foot width compared to baseline visit
Change in Swelling at Foot, Ankle & Mid-Calf (Circumference) | 6 weeks and 4 months post Lapiplasty® Procedure
  Change in swelling as compared to 0-2 week visit
Change in Scar Quality as Measured by Patient and Observer Scar Assessment Scale (POSAS) | 4 months, 6 months, and 12 months post Lapiplasty® Procedure
  Change in scar quality in comparison to baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Jody McAleer, DPM, FACFAS, Principal Investigator — JCMG - Podiatry
Locations (10):
- United States (10):
  - DOC - Decatur Orthopaedic Clinic, Decatur, Alabama
  - DOC - Decatur Orthopaedic Clinic, Hartselle, Alabama
  - Phoenix Foot and Ankle Institute, Scottsdale, Arizona
  - Orlando Foot and Ankle Clinic - Waterford Lakes Office, Orlando, Florida
  - JCMG - Podiatry, Jefferson City, Missouri
  - Desert Orthopaedic Center, Las Vegas, Nevada
  - University of Pennsylvania / Penn Medicine, Philadelphia, Pennsylvania
  - Stonebriar Foot and Ankle, Frisco, Texas
  - Foot & Ankle Associates of North Texas - Keller, Keller, Texas
  - Sports Medicine Associates of San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No